CLINICAL TRIAL: NCT04623710
Title: A Phase 1, Open-Label, Multiple-Dose, Parallel Study to Determine the Effect of Renal Impairment on the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of ALXN2050 in Adult Participants
Brief Title: Study of ALXN2050 in Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-108
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Renal Impairment; Healthy
Keywords: Factor D Inhibitor; Pharmacokinetics; Pharmacodynamics; Safety; ALXN2050
MeSH Terms: conditions — Renal Insufficiency | interventions — rhoA GTP-Binding Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Severe Impaired Renal Function (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050
- Cohort 2: Moderate Impaired Renal Function (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050
- Cohort 3: Mild Impaired Renal Function (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050
- Cohort 4: Healthy Control (Experimental): Participants will receive ALXN2050.
  Interventions: Drug: ALXN2050

INTERVENTIONS:
Drug: ALXN2050 — ALXN2050 (120 milligrams) will be administered orally twice daily on Days 1 through 3, with an additional dose (120 milligrams) administered orally on the morning of Day 4.
  Other Names: ACH-0145228 (formerly)

SUMMARY:
This study will investigate the impact of impaired renal function on the plasma pharmacokinetics of ALXN2050 in order to provide dosing recommendations for future indications in individuals with impaired renal function.

DETAILED DESCRIPTION:
The study will initiate (Part 1) with participants with severe impaired renal function (Cohort 1) and their matched healthy control participants (Cohort 4). Following data review, the study may proceed (Part 2) with participants with moderate (Cohort 2) and mild (Cohort 3) impaired renal function if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight must be at least 50.0 kilograms (kg) and body mass index (BMI) within the range of 18.0 - 40.0 kg/meter squared (m^2) (inclusive) at the time of signing the informed consent.
2. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
3. Must agree to receive prophylactic antibiotics to mitigate the potential risk of meningococcal infection.

   Participants with Impaired Renal Function
4. Aside from impaired renal function, sufficiently healthy for study participation based upon medical history, physical examination, neurological examination, laboratory tests, vital signs, and electrocardiograms (ECGs).
5. A clinical diagnosis of impaired stable renal function.
6. No clinically significant change in renal status at least 1 month prior to first dose of study intervention and is not currently or has not previously been on hemodialysis or did not have any history of peritoneal dialysis.
7. Stable creatinine clearance.
8. Must be on a stable medication regimen. Concomitant medications must be approved by Alexion unless presented in the list of common concurrent medications for participants with impaired renal function.

   Matched Healthy Control Participants with Normal Renal Function
9. Must match the sex and the race (similar ratio of white and non-white) of participants with impaired renal function, and at screening, age must be within ± 10 years and BMI must be within ± 20% of the matching participants with impaired renal function
10. Healthy as determined by medical evaluation, including medical history, physical examination, neurological examination, laboratory tests, vital signs, and ECGs, and who possess a baseline eGFR ≥ 90 mL/min/1.73 m^2, based on MDRD equation at screening.

Exclusion Criteria:

1. History or presence of seizures, head injury, head trauma, or any other brain disorder.
2. History of procedures that could alter absorption or excretion of orally administered drugs.
3. History of meningococcal infection or a first-degree relative with a history of meningococcal infection.
4. Body temperature ≥38.0°Celcius at screening or check-in or history of febrile illness or other evidence of infection, systemic or otherwise, within 14 days prior to the first dose of study intervention.
5. Participants with CH50 results outside the reference ranges at screening, unless approved by Alexion
6. Significant blood loss or donation of blood within 3 months prior to the first dose of study intervention, donation of plasma within 30 days prior to the first dose of study intervention, receipt of blood products within 6 months prior to first dose of study intervention, or receipt of a vaccine within 30 days prior to the first dose of study intervention.
7. Current enrollment or past participation within the last 30 days (or 5 half-lives, whichever is longer) prior to the first dose of study intervention in the current clinical study or any other clinical study involving an investigational study intervention or any other type of medical research.
8. History or presence of drug or alcohol abuse within 1 year prior to the first dose of study intervention, current tobacco user, or positive results for alcohol and/or drug screen at screening or check-in.
9. Pregnant or lactating.
10. Does not produce sufficient urine output to permit urine sampling at screening and/or check-in or has a history of urinary incontinence prior to check-in.
11. History of kidney transplant or actively on a transplant waiting list prior to check-in.
12. Any acute or chronic non-renal condition prior to check-in that would limit the participant's ability to complete or participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Area Under The Concentration-time Curve From Time 0 To The 12-hour Time Point (AUC0-12) Of Plasma ALXN2050 After Steady-state | Up to 72 hours postdose
Area Under The Concentration-time Curve Calculated To The Last Observable Concentration At Time t (AUCt) Of Plasma ALXN2050 After Steady-state | Up to 72 hours postdose
Maximum (Peak) Steady-state Plasma Concentration (Cmax,ss) Of Plasma ALXN2050 | Up to 72 hours postdose
Time To Reach Maximum (Peak) Plasma Concentration Following ALXN2050 Administration At Steady-state (Tmax,ss) | Up to 72 hours postdose

SECONDARY OUTCOMES:
Change From Baseline In Complement Factor D Concentration At 24, 48, And 72 Hours Postdose | Baseline, 24, 48, and 72 hours postdose
Change From Baseline In Plasma b Fragment Of Complement Factor B Concentration | Baseline, up to 72 hours postdose
Change From Baseline In Complement Alternative Pathway Activity | Baseline, up to 72 hours postdose
Number Of Participants Receiving ALXN2050 With Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up (30 [+/- 2] days after last study drug administration)]

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Trial Site, Hialeah, Florida
  - Clinical Trial Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No